CLINICAL TRIAL: NCT05094856
Title: Effects of Fluid Therapy on Peripheral TIssue Perfusion During Sepsis/Septic Shock
Brief Title: Effects of Fluid Therapy on Peripheral TIssse Perfusion During Sepsis/Septic Shock
Acronym: REPTILOS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Grifols (funder) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP210918
Record Dates: First submitted 2021-07-31; First posted 2021-10-26 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock; Sepsis
Keywords: Endothelial dysfunction; Albumin; Fluid Therapy; Peripheral Tissue Perfusion; Septic shock; Microcirculatory effects; Hemodynamic effects; sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Effect of volume expansion by albumin on the correction of peripheral tissue hypoperfusion: Effect of volume expansion by albumin on the correction of peripheral tissue hypoperfusion by measuring the proportion of patients who normalized their cutaneous re-coloring time (CRT) measured at the index level, defined by a value <3 seconds at H1. The clinical measurement method has been standardized in the participating departments and has been used for several years in clinical practice.
- Effect of volume expansion by saline on the correction of peripheral tissue hypoperfusion: Effect of volume expansion by saline on the correction of peripheral tissue hypoperfusion by measuring the proportion of patients who normalized their cutaneous re-coloring time (CRT) measured at the index level, defined by a value <3 seconds at H1. The clinical measurement method has been standardized in the participating departments and has been used for several years in clinical practice.

SUMMARY:
Compare the effect of volume expansion by saline versus albumin on the correction of peripheral tissue hypoperfusion by measuring Index skin recoloration time (CRT) at H0 and H1

DETAILED DESCRIPTION:
This is a transversal study allowing to compare the effect of volume expansion by saline versus albumin on the correction of peripheral tissue hypoperfusion

Design:

• A multicentric, open-label, transversal study

Sample size :

60 patients

Assessement:

Between the admission to intensive care and 48 hours after admission, the patient will be included after collection of the non-opposition form.

The patient will receive volume expansion either by 0.9% saline (500mL) or by 20% albumin (100mL) over 15 minutes.

Repeated clinical measurements will be performed at H0, H0.5 and H1 (respectively at 0, 30 and 60 minutes).

A blood sample will be taken just before the volume expansion and 4 hours after, at the same time as the samples usually taken as part of the treatment.

No interim analysis is planned. Analysis will be performed at the end of the study after data review and freezing of data base.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Sepsis or
* Septic shock within 24 hours of admission to intensive care with a stable dose of norepinephrine for at least 2 hours to maintain MAP> 65mmHg
* CRT index> 3 seconds despite the initial resuscitation (administration of antibiotics, volume expansion by crystalloids of 20 mL / Kg, noradrenaline started) between the admission to intensive care and H48 from admission to intensive care
* Non-opposition of the patient collected by the doctor in charge of the patient between H0 and H6 after admission if the patient is vigilant, otherwise a procedure for collecting non-opposition from relatives will be carried out with collection of the non-opposition of the patient once he is able to give it.
* Affiliation to a social security regimen (excluding AME)

Exclusion Criteria:

* Patient COVID-19 (+) with respiratory impairment
* Pregnant and lactating woman
* Patient under Guardianship / Curatorship
* Refusal to participate
* CRT not evaluable (dark or damaged skin)
* Moribund patient
* Estimated life expectancy less than 1 month
* Participation in another interventional research involving the human person or period of exclusion at the end of a previous research involving the human person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis/septic shock hospitalized in intensive care with signs of peripheral hypoperfusion persisting despite the initial resuscitation.
  Septic shock corresponds to patients with sepsis (infection + 2 SOFA points according to the latest international definition and the need to administer noradrenaline to maintain mean arterial pressure> 65 mmHg.
  In total, patients with reanimated and hemodynamically stabilized sepsis/septic shock will be included. The diagnostic and therapeutic management will comply in all points with the usual service protocol and international recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Compare the effect of volume expansion by saline versus albumin on the correction of peripheral tissue hypoperfusion by measuring Index skin recoloration time (CRT) at H0 and H1 | 1 hour
  Proportion of patients who normalized their cutaneous re-coloring time (CRT) measured at the index level, defined by a value <3 seconds at H1. The clinical measurement method has been standardized in the participating departments and has been used for several years in clinical practice.

SECONDARY OUTCOMES:
CRT Measure | 4 hours
  Clinical tissue perfusion parameters will be measured clinically every 30 minutes, as usual in patients with septis/septic shock.
mottling score measure | 4 hours
  Clinical tissue perfusion parameters will be measured clinically every 30 minutes, as usual in patients with sepsis/septic shock.
Diuresis | 4 hours
  Clinical tissue perfusion parameters will be measured clinically every 30 minutes, as usual in patients with sepsis/septic shock.
Variations in cardiac flow | 4 hours
  Clinical tissue perfusion parameters will be measured clinically every 30 minutes, as usual in patients with sepsis/septic shock.
Variations in the biological parameters | 4 hours
  Variations in the biological parameters between H0 and H4 will be analyzed from 5 ml of blood taken in addition, in accordance with the usual practice, in a sepsis/septic shock:
  * IL-6, IL-1b, Il-8, TNFa, IL-10
  * Syndecan-1, heparan sulfat, hyaluronat
  * Circulating microparticles

CONTACTS AND LOCATIONS:
Overall Officials: Hafid AIT-OUFELLA, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gabarre P, Desnos C, Morin A, Missri L, Urbina T, Bonny V, Turpin M, Baudel JL, Berard L, Montil M, Guidet B, Voiriot G, Joffre J, Maury E, Ait-Oufella H. Albumin versus saline infusion for sepsis-related peripheral tissue hypoperfusion: a proof-of-concept prospective study. Crit Care. 2024 Feb 7;28(1):43. doi: 10.1186/s13054-024-04827-0. PMID 38326920